CLINICAL TRIAL: NCT00848289
Title: Genetic Susceptibility to Bladder Cancer: A Molecular Epidemiology Approach
Brief Title: Genetic Susceptibility to Bladder Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LAB98-040; LAB98-040 (Other: MD Anderson Cancer Center); 5P50CA091846-14 (NIH); H-8577 (Other: Baylor College of Medicine); 5R01CA074880 (NIH); NCI-2021-06405 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Genetic susceptibility; Increased Risk
MeSH Terms: conditions — Urinary Bladder Neoplasms; Genetic Predisposition to Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood (about 40 cc or 8 teaspoons), urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Bladder Cancer: Patients diagnosed with superficial or muscle-invasive bladder cancer. Specimens, personal and follow-up telephone interviews will be collected and conducted.
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Interviews — Data collected by personal interview for Epidemiology and Nutrition Questionnaires, with personal and follow-up telephone interviews.

SUMMARY:
This clinical research study will identify biologic and lifestyle factors which increase a person's risk of developing specific cancer. Researchers propose to conduct a case-control study examining interindividual differences in susceptibility to tobacco carcinogenesis as predictors of bladder cancer risk. We will measure susceptibility to tobacco carcinogenesis and this will include studies of the genetic modulation of carcinogen activation and detoxification and of chromosome sensitivity to tobacco mutagens.

DETAILED DESCRIPTION:
Researchers propose to conduct a case-control study examining interindividual differences in susceptibility to tobacco carcinogenesis as predictors of bladder cancer risk. We will measure susceptibility to tobacco carcinogenesis and this will include studies of the genetic modulation of carcinogen activation and detoxification and of chromosome sensitivity to tobacco mutagens.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a histologically confirmed diagnosis of superficial or muscle-invasive bladder cancer
* Subject is a Texas resident.
* Subject can understand English or a qualified translator is available for the interview.
* Subjects of any age, gender, or ethnicity are eligible to participate in the study.
* Subject consents to participate in the study.

Exclusion Criteria:

* Subject has had prior treatment with systemic chemotherapy or radiotherapy in the past 6 months.
* Subject has been diagnosed with superficial or muscle-invasive bladder cancer more than twelve months ago.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who have been diagnosed with bladder cancer or who is healthy is eligible to participate without regard to age, sex, or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 6086 (Actual)
Dates: Start 1998-02-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of mutagen sensitivity susceptibility assays that quantifies the number of lymphocytic chromatid breaks induced by in vitro exposure to bleomycin and the number of breaks induced by in vitro exposure to a tobacco carcinogen | After last subject has completed the study, up to 5 years
  Mutagen sensitivity as measured by quantifying the number of lymphocytic chromatid breaks and comet tail moments induced by in vitro exposure to bleomycin (a radiomimetic agent) and benzo[a]pyrene diol epoxide (BPDE, a tobacco carcinogen) in bladder cancer cases in comparison to data for controls

SECONDARY OUTCOMES:
Frequencies of polymorphisms in those genes that regulate the metabolism of carcinogens in tobacco smoke | After the last subject completes the study, up to 5 years
Associations between the cytogenetic, molecular components and epidemiologic covariates (age, sex, ethnicity, cigarette smoking status, alcohol use, dietary intake, and family history of cancer) in risk of bladder cancer | After the last subject has completed the study, up to 5 years per individual participation

CONTACTS AND LOCATIONS:
Overall Officials: Jian Gu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org